CLINICAL TRIAL: NCT04236544
Title: Impact of a Multimedia Website With Patient Experiences of Multiple Sclerosis (PExMS) on Immunotherapy Decision-making: a Pilot Randomised Controlled Trial in a Mixed-methods Design
Brief Title: Patient Experiences of Multiple Sclerosis (PExMS)
Acronym: PExMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Marianne-Strauss-Klinik, Berg, Germany (Unknown); Gesundheitszentrum St. Johannes Hospital, Bonn, Germany (Unknown); University Hospital Cologne, Cologne, Germany (Unknown); Rechts der Isar Hospital, Munich, Germany (Unknown); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PExMS
Record Dates: First submitted 2019-12-06; First posted 2020-01-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Patient Engagement; Self Efficacy
Keywords: multiple sclerosis; decision making; decision support; web-based experiential information; patient experiences; narrative information
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Patient Participation

STUDY DESIGN:
Intervention Model Description: After informed consent, baseline data will be obtained by the staff member responsible for enrolment and people with multiple sclerosis will be randomly allocated in blocks with variable block length at a 1:1 ratio to the intervention or the control group. The allocation sequence will be computer-generated by a statistician not involved in the conduction of the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We will explain in our information and consent form that we intend to assess whether patients with mutiple sclerosis find different health information websites helpful on a range of self-reported outcomes. Researchers involved in study recruitment, administration of interventions and data analysis will be blind to the allocation of intervention and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PExMS and DECIMS-Wiki (Experimental): After allocation, the intervention group will receive access via a data-protected study platform (www.erecover.de) to PExMS and DECIMS-Wiki for a two-week period. The former is a multimedia website providing experiential information. DECIMS (Decision coaching in MS)-Wiki (www.wiki2.kkn-ms.de) is an evidence-based patient information website focusing multiple sclerosis immunotherapies. Afterwards, primary and secondary outcome measures will be obtained. In a next step, patient will be asked for their treatment decision in a physician encounter.
  Interventions: Behavioral: PExMS and DECIMS-Wiki
- DECIMS-Wiki (Active Comparator): After allocation, the control group will receive access to the DECIMS-Wiki for a two-week period. DECIMS (Decision coaching in MS)-Wiki (www.wiki2.kkn-ms.de) is an evidence-based patient information website focusing multiple sclerosis immunotherapies. Afterwards, primary and secondary outcome measures will be obtained. In a next step, patient will be asked for their treatment decision in a physician encounter.
  Interventions: Behavioral: DECIMS-Wiki

INTERVENTIONS:
Behavioral: PExMS and DECIMS-Wiki — The intervention consists of an information provision on immunotherapies as a combination of factual and experiential information. PExMS is a multimedia website providing patient experiences with MS in everyday life and with therapies illustrated by video, audio and text files of 48 persons with multiple sclerosis. The development of the intervention followed largely recommendation for standardised qualitative research provided by international DIPEx (Database of Individual Patients' Experience of illness) association, which use standardised qualitative research methods to provide 'balanced' information from original interview data. Data for the website was generated in a qualitative interview study with relapsing remitting multiple sclerosis patients across Germany. DECIMS (Decision coaching in MS)-Wiki (www.wiki2.kkn-ms.de) is an evidence-based patient information website focusing multiple sclerosis immunotherapies.
  Arms: PExMS and DECIMS-Wiki
Behavioral: DECIMS-Wiki — The active comparator is DECIMS-Wiki, which is an evidence-based online information platform. It is considered to be excellent factual information about immunotherapies for multiple sclerosis.
  Arms: DECIMS-Wiki

SUMMARY:
Besides coping with the diagnosis, people with multiple sclerosis have to make complex decisions such as deciding about immunotherapies. They search not only for factual information, but also for reports of patient experiences (PEx). The investigators aim to evaluate in a randomised controlled pilot trial whether a website presenting PEx as an adjunct to factual information may help people with multiple sclerosis in their immunotherapy decision-making processes.

DETAILED DESCRIPTION:
A variety of management options (e.g. immunotherapies, lifestyle interventions, and rehabilitation) are available for people with relapsing-remitting multiple sclerosis. Besides coping with the diagnosis, people with multiple sclerosis have to make complex decisions such as deciding about immunotherapies. In addition to factual information, reports of patient experiences (PEx) may support patients in decision-making. The added value of PEx in decision-making is not clear and controlled studies are rare. Therefore, systematic methods are necessary in order to develop and analyse PEx. As there are no evaluated PEx for multiple sclerosis in Germany, the investigators are currently creating a website presenting PEx structured according to topics and illustrated by video, audio and text files.

The investigators aim to evaluate whether PEx may help people with multiple sclerosis in their immunotherapy decision-making processes.

This project will follow the Medical Research Council framework for development and evaluation of complex interventions. After the development of a website with PEx, a randomised controlled pilot trial will be conducted in five neurological practices/clinics including 55 people with relapsing-remitting multiple sclerosis and accompanied by a process evaluation.

Participants will be randomly assigned either to i) an intervention group with a two weeks access to an evidence-based patient information resource and the PExMS-website as an adjunct or to ii) the control group with access to evidence information alone.

A 6-members advisory panel involving representatives of people with multiple sclerosis, researchers, and neurologists, who accompany the whole project will mentor this pilot RCT. The ethical committee of the Hamburg Chamber of Physicians approved the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* persons with relapsing-remitting multiple sclerosis
* being ≥18 years old
* considering starting, switching or stopping any immunotherapy

Exclusion Criteria:

* persons with secondary progressive multiple sclerosis or primary progressive multiple sclerosis
* persons with major cognitive deficits
* persons having poor German language skills
* persons who participated in the development phase of the PExMS-website, which took place prior to the pilot randomised controlled trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Testing the feasibility of an intervention using patients' experiences as a supplement to evidence-based information in a pilot randomized controlled trial | Baseline and up to 6 months after beginning, changing or stopping of the immunotherapy
  The specific measures to test the feasibility are:
  * Number of participants consented, recruited, randomized, withdrawn, and retained
  * Numbers of participants with completed outcome measures or lost to follow-up
  * Acceptability of the intervention in terms of site visits, frequency, and duration of usage as well as experience, barriers, and facilitators to use the intervention - from persons with MS and health professionals from participating study centers
  * Acceptability of the study procedures in terms of barriers and facilitators to implementation - from persons with MS and participating study centers.

SECONDARY OUTCOMES:
Preparation for Decision Making | Up to 14 days after usage of intervention or comparator website(s)
  To assess how useful a decision support intervention is in preparing patients with multiple sclerosis to communicate at a consultation visit and making a decision concerning a therapy, the 10-item Preparation for Decision Making (PrepDM) scale will be used. It has a five-point-Likert scale format and is designed to be administered after the consultation visit to discuss treatment options. Higher scores show a higher perceived level of preparation for decision-making.
Decisional Conflict | Baseline and up to 14 days after usage of intervention or comparator website(s)
  The 4-item yes/no response "Sure of myself, Understand information, Risk-benefit ratio, Encouragement" (SURE) screening test addresses decisional conflict in patients. This screening instrument was developed to help health professionals assess patients' perception of uncertainty about decision-making for a therapy. The SURE screening test has dichotomous questions, where "yes" equals 1 point and "no" equals 0 point. If the total score is less than 4, it indicates the probability that the patient experiences clinically significant decisional conflict.
Self-reported impact of eHealth on its users | eHIQ-Part-1 at baseline and the eHIQ-Part-2 up to 14 days after usage of intervention or comparator website(s)
  The eHealth Impact Questionnaire (eHIQ) measures users' attitudes towards a website which they recently viewed. It is divided into the 11-item eHIQ-Part 1, asking for general attitudes towards using the internet to access health information and the 26-item eHIQ-Part 2, which is related to the effects of using a specific health-related website on three subscales: 1) confidence and identification, 2) information and presentation and 3) understanding and motivation. Both answering formats range from 1 (strongly disagree) to 5 (strongly agree). Moreover, identifying with others who show their experiences on a website, knowing that other pwMS are handling similar problems and learning how they manage difficult issues can reduce the feeling of isolation and improve the sense of social support. Reformulated items from the subscale "confidence and identification" of the eHIQ will be used to assess social support.
Affective forecasting in regard to immunotherapies | Baseline and up to 14 days after usage of intervention or comparator website(s) and and 6 months after the beginning of the immunotherapy
  As suitable instruments to assess affective forecasts regarding the use of immunotherapies were lacking, we developed the 'Affective Forecasting in Immunotherapy for Multiple Sclerosis questionnaire' (AForT-MS). It consists of items addressing anticipated positive and negative emotions, fears and hopes, regret, and focalism in regard to immunotherapies. Ratings have to be performed based on a 6-point Likert scale. Cognitive interviews with n=6 persons with MS were executed using the verbal probing method to identify potentially problematic questions, difficulties and ambiguities which could lead to unintended answers and to improve the questionnaire. The online version of the AFort-MS will be tested in a sample of persons with MS being in the decision-making process to start, change or stop an immunotherapy and revised afterwards. In a second step, we will administer the revised AForT-MS to the same sample of persons with MS in the pilot RCT to conduct an exploratory factor analysis.
Self-confidence in decision-making | Baseline and up to 14 days after usage of intervention or comparator website(s)
  The 11-item Decision Self-Efficacy Scale (DSES) measures self-confidence in decision-making on a five-point-Likert scale. It ranges between 0 (not at all confident) and 4 (very confident). For the total score, items are summed, divided by 11 and multiplied by 25. A total score of 0 means 'extremely low self-efficacy' and a score of 100 means 'extremely high self-efficacy'.
Patients' beliefs about the necessity of their medication and their concerns about the current medication | Baseline and up to 14 days after usage of intervention or comparator website(s)
  The 11-item subscale 'Specific Necessity Beliefs' of the 'Beliefs about Medicines Questionnaire' (BMQ) assesses specific concerns about the current medication. All items are scored on a 5-point Likert-scale, ranging from "0" (totally disagree) to "4" (totally agree). Scores obtained for individual items are summed. Higher scores indicate stronger beliefs.
Adherence | 6 months after beginning, changing or stopping of the immunotherapy
  Patients who belief in a strong necessity of their medication have higher adherence behavior. We hypothesize that patients' experiences about the aspects of an immunotherapy in everyday life may prepare other persons with MS for difficulties they might face and improve their resilience under this condition and the adherence to a given immunotherapy.
  Participants have to answer adherence questions referred to the last four weeks for oral DMTs and self-injectables or the past six months for taking infusions.

OTHER OUTCOMES:
Symptoms of Anxiety and Depression | Baseline and up to 14 days after usage of intervention or comparator website(s)
  As a control parameter, the Hospital Anxiety and Depression Scale (HADS) will be administered. Seven of the items relate to anxiety and seven relate to depression. Each item on the HADS is scored from 0-3 and this means that a person with multiple sclerosis can score between 0 and 21 for either anxiety or depression. A score of 0-7 means 'Normal', 8-10 means 'Borderline abnormal' and 11-21 means 'Abnormal'.
Patient-reported disability | Baseline
  The Patient Determined Disease Steps (PDDS) measures patient-reported disability of persons with multiple sclerosis. The PDDS has nine ordinal levels ranging between 0 (normal) and 8 (bedridden).
Stage of Decision Making | Baseline
  The 'Stage of Decision Making' questionnaire asks for the patient's readiness to engage in decision-making, progress in decision-making and susceptibility to considering or re-considering options. It may be useful in screening out persons with multiple sclerosis who may not benefit from decision aids interventions.
Control Preferences for involvement in treatment decisions | Baseline and up to 14 days after usage of intervention or comparator website(s)
  The 5-item Control Preferences Scale (CPS) assess patients' preferences for involvement in treatment decisions. It consists of five ''cards'' on a board, each illustrating a different role in decision-making by means of a cartoon and short descriptive statement. The examiner asks the respondent to choose the preferred card, which is then covered up and cannot be chosen again. Afterwards, the examiner asks the respondent to choose the preferred card from the remaining four cards. The procedure continues until one card is left. If the second preference is incongruent with the first, the test is immediately re-administered. Six scores are possible based on the subject's two most preferred roles: active-active, active-collaborative, collaborative-active, collaborative-passive, passive-collaborative and passive-passive.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

IPD SHARING:
Plan to Share IPD: Yes
The study centre will coordinate the intra-study data sharing process publishing anonymized data set in major journals. The results of our study will be presented at national and international conferences and published in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will become available when summary data are published.
Access Criteria: IPD will be shared upon request from the principal investigator.

REFERENCES:
- [Background] Browne P, Chandraratna D, Angood C, Tremlett H, Baker C, Taylor BV, Thompson AJ. Atlas of Multiple Sclerosis 2013: A growing global problem with widespread inequity. Neurology. 2014 Sep 9;83(11):1022-4. doi: 10.1212/WNL.0000000000000768. No abstract available. PMID 25200713
- [Background] WHO. Atlas multiple sclerosis resources in the world 2008. Geneva; London: World Health Organization; Multiple Sclerosis International Federation; 2008. 51 p.
- [Background] Heesen C, Kasper J, Segal J, Kopke S, Muhlhauser I. Decisional role preferences, risk knowledge and information interests in patients with multiple sclerosis. Mult Scler. 2004 Dec;10(6):643-50. doi: 10.1191/1352458504ms1112oa. PMID 15584489
- [Background] Heesen C, Schaffler N, Kasper J, Muhlhauser I, Kopke S. Suspected multiple sclerosis - what to do? Evaluation of a patient information leaflet. Mult Scler. 2009 Sep;15(9):1103-12. doi: 10.1177/1352458509106508. Epub 2009 Jul 22. PMID 19625332
- [Background] Heesen C, Kolbeck J, Gold SM, Schulz H, Schulz KH. Delivering the diagnosis of MS--results of a survey among patients and neurologists. Acta Neurol Scand. 2003 May;107(5):363-8. doi: 10.1034/j.1600-0404.2003.00086.x. PMID 12713529
- [Background] Rahn AC, Kopke S, Kasper J, Vettorazzi E, Muhlhauser I, Heesen C. Evaluator-blinded trial evaluating nurse-led immunotherapy DEcision Coaching In persons with relapsing-remitting Multiple Sclerosis (DECIMS) and accompanying process evaluation: study protocol for a cluster randomised controlled trial. Trials. 2015 Mar 21;16:106. doi: 10.1186/s13063-015-0611-7. PMID 25872529
- [Background] Newhouse N, Martin A, Jawad S, Yu LM, Davoudianfar M, Locock L, Ziebland S, Powell J. Randomised feasibility study of a novel experience-based internet intervention to support self-management in chronic asthma. BMJ Open. 2016 Dec 28;6(12):e013401. doi: 10.1136/bmjopen-2016-013401. PMID 28031210
- [Background] Ziebland S, Powell J, Briggs P, Jenkinson C, Wyke S, Sillence E, Harris P, Perera R, Mazanderani F, Martin A, Locock L, Kelly L, Booth M, Gann B, Newhouse N, Farmer A. Examining the role of patients' experiences as a resource for choice and decision-making in health care: a creative, interdisciplinary mixed-method study in digital health. Southampton (UK): NIHR Journals Library; 2016 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK401199/ PMID 27929620
- [Background] Powell J, Newhouse N, Martin A, Jawad S, Yu LM, Davoudianfar M, Locock L, Ziebland S. A novel experience-based internet intervention for smoking cessation: feasibility randomised controlled trial. BMC Public Health. 2016 Nov 11;16(1):1156. doi: 10.1186/s12889-016-3821-3. PMID 27835953
- [Background] Dillard AJ, Fagerlin A, Dal Cin S, Zikmund-Fisher BJ, Ubel PA. Narratives that address affective forecasting errors reduce perceived barriers to colorectal cancer screening. Soc Sci Med. 2010 Jul;71(1):45-52. doi: 10.1016/j.socscimed.2010.02.038. Epub 2010 Mar 21. PMID 20417005
- [Background] Bekker HL, Winterbottom AE, Butow P, Dillard AJ, Feldman-Stewart D, Fowler FJ, Jibaja-Weiss ML, Shaffer VA, Volk RJ. Do personal stories make patient decision aids more effective? A critical review of theory and evidence. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S9. doi: 10.1186/1472-6947-13-S2-S9. Epub 2013 Nov 29. PMID 24625283
- [Background] Engler J, Adami S, Adam Y, Keller B, Repke T, Fugemann H, Lucius-Hoene G, Muller-Nordhorn J, Holmberg C. Using others' experiences. Cancer patients' expectations and navigation of a website providing narratives on prostate, breast and colorectal cancer. Patient Educ Couns. 2016 Aug;99(8):1325-32. doi: 10.1016/j.pec.2016.03.015. Epub 2016 Mar 17. PMID 27067064
- [Background] Entwistle VA, France EF, Wyke S, Jepson R, Hunt K, Ziebland S, Thompson A. How information about other people's personal experiences can help with healthcare decision-making: a qualitative study. Patient Educ Couns. 2011 Dec;85(3):e291-8. doi: 10.1016/j.pec.2011.05.014. Epub 2011 Jun 8. PMID 21652162
- [Background] Giesler JM, Keller B, Repke T, Leonhart R, Weis J, Muckelbauer R, Rieckmann N, Muller-Nordhorn J, Lucius-Hoene G, Holmberg C. Effect of a Website That Presents Patients' Experiences on Self-Efficacy and Patient Competence of Colorectal Cancer Patients: Web-Based Randomized Controlled Trial. J Med Internet Res. 2017 Oct 13;19(10):e334. doi: 10.2196/jmir.7639. PMID 29030329
- [Background] Shaffer VA, Zikmund-Fisher BJ. All stories are not alike: a purpose-, content-, and valence-based taxonomy of patient narratives in decision aids. Med Decis Making. 2013 Jan;33(1):4-13. doi: 10.1177/0272989X12463266. Epub 2012 Oct 11. PMID 23065418
- [Background] Winterbottom A, Bekker HL, Conner M, Mooney A. Does narrative information bias individual's decision making? A systematic review. Soc Sci Med. 2008 Dec;67(12):2079-88. doi: 10.1016/j.socscimed.2008.09.037. Epub 2008 Oct 24. PMID 18951673
- [Background] Graham ID OCA. User Manual - Preparation for Decision Making Scale. In: Institute OHR, editor. Ottawa1995.
- [Background] Rahn AC, Kopke S, Backhus I, Kasper J, Anger K, Untiedt B, Alegiani A, Kleiter I, Muhlhauser I, Heesen C. Nurse-led immunotreatment DEcision Coaching In people with Multiple Sclerosis (DECIMS) - Feasibility testing, pilot randomised controlled trial and mixed methods process evaluation. Int J Nurs Stud. 2018 Feb;78:26-36. doi: 10.1016/j.ijnurstu.2017.08.011. Epub 2017 Aug 26. PMID 28982479
- [Background] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Background] Heesen C, Kasper J, Fischer K, Kopke S, Rahn A, Backhus I, Poettgen J, Vahter L, Drulovic J, Van Nunen A, Beckmann Y, Liethmann K, Giordano A, Fulcher G, Solari A; AutoMS-group. Risk Knowledge in Relapsing Multiple Sclerosis (RIKNO 1.0)--Development of an Outcome Instrument for Educational Interventions. PLoS One. 2015 Oct 2;10(10):e0138364. doi: 10.1371/journal.pone.0138364. eCollection 2015. PMID 26430887
- [Background] Heesen C, Pottgen J, Rahn AC, Liethmann K, Kasper J, Vahter L, Drulovic J, Van Nunen A, Wilkie D, Beckmann Y, Paul F, Kopke S, Giordano A, Solari A; AutoMS-group. What should a person with relapsing-remitting multiple sclerosis know? - Focus group and survey data of a risk knowledge questionnaire (RIKNO 2.0). Mult Scler Relat Disord. 2017 Nov;18:186-195. doi: 10.1016/j.msard.2017.09.020. Epub 2017 Sep 21. PMID 29141808
- [Background] Marteau TM, Dormandy E, Michie S. A measure of informed choice. Health Expect. 2001 Jun;4(2):99-108. doi: 10.1046/j.1369-6513.2001.00140.x. PMID 11359540
- [Background] Kopke S, Kasper J, Flachenecker P, Meissner H, Brandt A, Hauptmann B, Bender G, Backhus I, Rahn AC, Pottgen J, Vettorazzi E, Heesen C. Patient education programme on immunotherapy in multiple sclerosis (PEPIMS): a controlled rater-blinded study. Clin Rehabil. 2017 Feb;31(2):250-261. doi: 10.1177/0269215516639734. Epub 2016 Jul 10. PMID 27072153
- [Background] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] De Las Cuevas C, Penate W. Validity of the Control Preferences Scale in patients with emotional disorders. Patient Prefer Adherence. 2016 Nov 15;10:2351-2356. doi: 10.2147/PPA.S122377. eCollection 2016. PMID 27895470
- [Background] Kelly L, Ziebland S, Jenkinson C. Measuring the effects of online health information: Scale validation for the e-Health Impact Questionnaire. Patient Educ Couns. 2015 Nov;98(11):1418-24. doi: 10.1016/j.pec.2015.06.008. Epub 2015 Jun 22. PMID 26162953
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Kelly L, Jenkinson C, Ziebland S. Measuring the effects of online health information for patients: item generation for an e-health impact questionnaire. Patient Educ Couns. 2013 Dec;93(3):433-8. doi: 10.1016/j.pec.2013.03.012. Epub 2013 Apr 15. PMID 23598293
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Learmonth YC, Motl RW, Sandroff BM, Pula JH, Cadavid D. Validation of patient determined disease steps (PDDS) scale scores in persons with multiple sclerosis. BMC Neurol. 2013 Apr 25;13:37. doi: 10.1186/1471-2377-13-37. PMID 23617555
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Derived] Barabasch A, Riemann-Lorenz K, Kofahl C, Scheiderbauer J, Eklund D, Kleiter I, Kasper J, Kopke S, Lezius S, Zapf A, Rahn AC, Heesen C. Impact of a multimedia website with patient experiences of multiple sclerosis (PExMS) on immunotherapy decision-making: study protocol for a pilot randomised controlled trial in a mixed-methods design. Pilot Feasibility Stud. 2021 Jan 7;7(1):16. doi: 10.1186/s40814-020-00749-0. PMID 33413658
- See also: O'Connor A. User Manual - Decision Self-Efficacy Scale 1995 — http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf
- See also: O'Connor AM. User Manual Stage of Decision Making 2003 — https://decisionaid.ohri.ca/docs/develop/Tools/Stage_Decision_Making_PAD.pdf